CLINICAL TRIAL: NCT01458899
Title: Phase I, Open-label, Randomized, Single-dose, Two Treatment (Fed Versus Fasted) Crossover Study to Assess the Effects of Food on the Pharmacokinetics of TC-5214 (S-Mecamylamine) in Healthy Subjects
Brief Title: Study in Healthy Subjects to Measure the Effects of Food on the Pharmacokinetics of TC-5214
Acronym: TC-5214
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4130C00025
Record Dates: First submitted 2011-10-17; First posted 2011-10-25 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Subjects
Keywords: Phase 1; healthy male; nonpregnant female; volunteers; pharmacokinetics; TC 5214; The effect of food on the pharmacokinetics of TC-5214

ARMS (2):
- A - first fed then fasted treatment (Experimental): TC-5214
  Interventions: Drug: TC-5214
- B - first fasted then fed treatment (Experimental): TC-5214
  Interventions: Drug: TC-5214

INTERVENTIONS:
Drug: TC-5214 — Oral tablets, single 4mg dose

SUMMARY:
(Food versus no food) crossover study to measure the effects of food on pharmacokinetics of TC-5214 (S-Mecamylamine) in healthy Subjects.

DETAILED DESCRIPTION:
Phase I, Open-label, Randomized, Single-dose, Two treatment (Fed Versus Fasted) Crossover Study to Assess the Effects of Food on the Pharmacokinetics of TC-5214 (S-Mecamylamine) in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written, and dated informed consent prior to any study specific procedures.
* Healthy male and nonpregnant, nonlactating female 18 to 55 years, inclusive, with suitable veins for cannulation or repeated venipuncture.
* Have a body mass index (BMI) between 19 and 32 kg/m2 and weigh at least 50 kg
* Be willing to eat the high-calorie, high-fat breakfast or fast accordingly
* Be able to understand and comply with the requirements of the study as judged by the Investigator

Exclusion Criteria:

* History of any clinically significant medical, neurologic, or psychiatric disease or disorder which, in the opinion of the Investigator and Sponsor, may either put the volunteer at risk because of participation in the study, or influence the results
* History of gastrointestinal surgery (except for appendectomy) or unintentional rapid weight loss
* History of seizure activity, including febrile seizures
* Past diagnosis of more than 1 episode of major depression
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
TC-5214 area under the plasma concentration time curve will be measured. | Pre dose, 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 7, 12, 24, 36, 48 and 72 hours post dose
TC-5214 maximum plasma concentration will be measured | Pre dose, 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 7, 12, 24, 36, 48 and 72 hours post dose

SECONDARY OUTCOMES:
The number of participants with adverse events | During day - 1, day 1, 2, 3 and 4 of treatment period
A change from baseline in laboratory assessments | During day - 1 and day 3 of visits 2 and 3 of treatment period
A change from baseline in vital signs | During day - 1, day 1, 2, 3 and 4 of treatment period
A change from baseline in physical examination | During day -1
Description of the pharmacokinetics (PK) of TC-5214 in terms of area under the curve over the time (AUC) and maximum concentration (Cmax) and terminal half-life | PK samles collected at pre dose, 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 7, 12, 24, 36, 48 and 72 hours post dose
Description of urine pharmacokinetics (PK) of TC-5214 in terms of the cumulative amount of drug excreted unchanged into urine from zero to time and renal clearance | PK samples collected at pre dose, 0 - 12, 12 - 24, 24 to 48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, Study Chair — AstraZeneca Kvambergagatan 12, 15185, Sodertalje, Sweden; David Mathews, MD, Principal Investigator — Quintiles, Inc. Overland Park US; Brendan Smyth, MD, Study Director — AstraZeneca 180 Concord Pike Wilmington, DE 19850-5437
Locations (1):
- Research Site, Overland Park, Kansas, United States